CLINICAL TRIAL: NCT00959972
Title: Varenicline Versus Transdermal Nicotine Patch for Smoking Cessation in Patients With Coronary Heart Disease: a Pilot Randomized Trial
Brief Title: Varenicline Versus Transdermal Nicotine Patch for Smoking Cessation in Patients With Coronary Heart Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Robert Reid, PhD, MBA, University of Ottawa Heart Insitute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIPRC-6551
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Coronary Heart Disease
Keywords: Varenicline; transdermal nicotine patch; cardiovascular disease; prevention; coronary heart disease; Smoking cessation
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases; Smoking Cessation | interventions — Varenicline; Tobacco Use Cessation Devices; Transdermal Patch; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Experimental): Participants randomized to varenicline will be administered 0.5 mg/day for 3 days, 0.5 mg twice daily for 4 days, then 1 mg twice daily thereafter for an additional 11 weeks.
  Interventions: Drug: Varenicline
- Transdermal Nicotine Patch (Experimental): Participants randomized to NRT will apply the patch immediately on the first day and each morning thereafter for 12 weeks. Doses of NRT will be 21 mg/day for the first 6 weeks, 14 mg/day for 4 weeks, then 7 mg/day for 2 weeks.
  Interventions: Drug: Transdermal Nicotine Patch

INTERVENTIONS:
Drug: Varenicline — Participants randomized to varenicline will be administered 0.5 mg/day for 3 days, 0.5 mg twice daily for 4 days, then 1 mg twice daily thereafter for an additional 11 weeks.
  Other Names: Champix; Chantix
  Arms: Varenicline
Drug: Transdermal Nicotine Patch — Participants randomized to NRT will apply the patch immediately on the first day and each morning thereafter for 12 weeks. Doses of NRT will be 21 mg/day for the first 6 weeks, 14 mg/day for 4 weeks, then 7 mg/day for 2 weeks.
  Other Names: Nicotine Patch; Patch; Nicoderm; NRT
  Arms: Transdermal Nicotine Patch

SUMMARY:
The purpose of this study is to determine if a new drug, varenicline, for smoking cessation is more effective than the standard nicotine replacement therapy aide currently used, "the patch" among smokers hospitalized with coronary heart disease.

DETAILED DESCRIPTION:
Quitting smoking is the single most effective intervention or treatment to reduce death rates in patients with coronary heart disease (CHD) who smoke. At the University of Ottawa Heart Institute (Ottawa, Canada), an institutional program is in place to ensure that staff consistently identify and document tobacco use status and treatment is offered to every smoker admitted to the Institute. Currently, nicotine replacement therapy (NRT) is the principal medication used in the program. Recently, a new medication, varenicline, was approved for smoking cessation in Canada. Varenicline appears be the most effective medication for cessation currently available. To date, most published studies of varenicline have been funded by the manufacturer and there are no published studies reporting how well it works in smokers hospitalized with heart disease.

This study involves sixty current smokers hospitalized at the UOHI for CHD. Consenting smokers will be randomly assigned to receive varenicline for 12 weeks or transdermal NRT for 12 weeks. Participants will also complete a two-page questionnaire inquiring about smoking history and previous attempts to quit, level of nicotine dependence, symptoms of nicotine withdrawal and self-efficacy with respect to quitting smoking. All participants will receive identical in-hospital counseling, self-help materials and follow-up support. The nurse specialists will also contact the participants by phone 3, 14, 30 and 50 days post-hospital discharge to check the patient's smoking status, assess the risk of relapse, and identify any adverse events that have occurred. The study will follow up with participants at 12 and 26 weeks post randomization asking about their smoking status (biochemically confirmed with a carbon monoxide monitor), adherence to prescribed medication, self-efficacy with respect to quitting smoking, nicotine withdrawal and smoking cessation resources used post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* smoking at least 10 cigarettes/day in the month prior to admission
* patient has been diagnosed with acute coronary syndrome (includes patients admitted for unstable angina or acute myocardial infarction), elective percutaneous coronary intervention, or coronary artery bypass surgery at any point in time
* motivated to stop smoking
* geographically available for follow-up visits (i.e., live within 1 hour of the study centre)

Exclusion Criteria:

* have been using NRT, Zyban (or Wellbutrin), and/or Champix for more than 72 hours
* have serious cardiac arrhythmias (e.g., tachycardia), vasospastic disease (e.g., Buerger's disease, Prinzmetal's variant angina)
* have severe renal impairment or are on dialysis
* unable to read and understand English
* patient is pregnant or breastfeeding or planning on becoming pregnant during the study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the biochemically confirmed (exhaled CO < 10 ppm) self-reported continuous abstinence for weeks 12 to 26. | 26 weeks

SECONDARY OUTCOMES:
Secondary outcomes will include adherence to prescribed pharmacotherapy measured at 12 weeks and measures of nicotine withdrawal and self-efficacy. | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Reid, PhD MBA, Principal Investigator — Ottawa Heart Institute Research Corporation; Andrew Pipe, MD, Study Chair — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Pipe A. Smoking. Can J Cardiol. 1999 Dec;15 Suppl G:77G-80G. No abstract available. PMID 10692663
- [Background] Critchley J, Capewell S. Smoking cessation for the secondary prevention of coronary heart disease. Cochrane Database Syst Rev. 2003;(4):CD003041. doi: 10.1002/14651858.CD003041. PMID 14583958
- [Background] Rigotti NA, Munafo MR, Stead LF. Interventions for smoking cessation in hospitalised patients. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD001837. doi: 10.1002/14651858.CD001837.pub2. PMID 17636688
- [Background] Reid RD, Pipe AL, Quinlan B. Promoting smoking cessation during hospitalization for coronary artery disease. Can J Cardiol. 2006 Jul;22(9):775-80. doi: 10.1016/s0828-282x(06)70294-x. PMID 16835672
- [Background] Meine TJ, Patel MR, Washam JB, Pappas PA, Jollis JG. Safety and effectiveness of transdermal nicotine patch in smokers admitted with acute coronary syndromes. Am J Cardiol. 2005 Apr 15;95(8):976-8. doi: 10.1016/j.amjcard.2004.12.039. PMID 15820167
- [Background] Gonzales D, Rennard SI, Nides M, Oncken C, Azoulay S, Billing CB, Watsky EJ, Gong J, Williams KE, Reeves KR; Varenicline Phase 3 Study Group. Varenicline, an alpha4beta2 nicotinic acetylcholine receptor partial agonist, vs sustained-release bupropion and placebo for smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):47-55. doi: 10.1001/jama.296.1.47. PMID 16820546
- [Background] Aubin HJ, Bobak A, Britton JR, Oncken C, Billing CB Jr, Gong J, Williams KE, Reeves KR. Varenicline versus transdermal nicotine patch for smoking cessation: results from a randomised open-label trial. Thorax. 2008 Aug;63(8):717-24. doi: 10.1136/thx.2007.090647. Epub 2008 Feb 8. PMID 18263663
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273